CLINICAL TRIAL: NCT06834919
Title: Translation, Cross-Cultural Adaptation, Validity and Reliability of Upper Limb Functional Index in Albanian Population
Brief Title: Upper Limb Functional Index
Acronym: ULFI-A
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jasemin Todri, Professor, Universidad Católica San Antonio de Murcia
Other Study IDs: 2456
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Upper Limb Function; Upper Limb Pain; Upper Limb; Injury, Superficial, Multiple; Upper Limb Rehabilitation
MeSH Terms: conditions — Wounds and Injuries | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational — Psychometric properties will be assessed by administering the questionnaire online to approximately 200 participants. Reliability will be estimated by assessing stability and homogeneity.

SUMMARY:
To translate and validate the Upper Limb Functional Index into Albanian for use in the Albanian-speaking population.

DETAILED DESCRIPTION:
The cross-cultural adaptation will be carried out in accordance with the internationally recommended methodology, following the guidelines: translation, back-translation; dissemination of questionnaires and data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain
* arm pain
* myofascial pain
* muscular pain
* trigger points
* arthritis

Exclusion Criteria:

* tumor
* metabolic disease
* neurologic conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants with myofascial pain.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-18 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Functional Index | 10 minutes
  The Upper Extremity Functional Index (ULFI) is a patient-reported outcome measure used to assess functional impairment in people with upper extremity musculoskeletal dysfunction. ULFI consists of 25 questions that assess the level of difficulty in performing activities of daily living using the upper extremities, including household and work activities, hobbies, lifting a bag of groceries, washing your scalp, pushing on your hands, driving, etc.